CLINICAL TRIAL: NCT02280551
Title: The Australian Parental Supply of Alcohol Longitudinal Study (APSALS)
Acronym: APSALS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Professor Richard P Mattick, Professor Richard P Mattick, The University of New South Wales
Other Study IDs: DP:1096668
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Alcohol Abuse
Keywords: adolescent; alcohol; parent; epidemiology
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adolescents: 1927 Grade 7 high school students
- Parent: A parent of each of the 1927 Grade 7 high school students

SUMMARY:
Parents can positively influence their children's alcohol use. One strategy they use is to provide their children with alcohol, believing it is the best way to teach their children how to drink responsibly. The impact of parental supply is not well understood and may be unintentionally harmful. This study will research the consequences of parental supply within the broader context of parent, child and peer relationships. It will help to determine how parental supply influences the different patterns of adolescent alcohol consumption over time, providing essential information to help parents prevent alcohol misuse in their children. Parents can play a pivotal role in prevention of alcohol misuse, but at present we don't know exactly how.

DETAILED DESCRIPTION:
Title: The Australian Parental Supply of Alcohol Longitudinal Study (APSALS): Can parents teach their children to drink alcohol responsibly? Or, is one drop a drop too many?

Background: The Australian Parental Supply of Alcohol Longitudinal Study (APSALS) was established to investigate the short- and long-term associations between exposure to parental alcohol provision, early adolescent alcohol initiation, subsequent alcohol use, and alcohol-related harms, controlling for a wide range of parental, child, familial, peer, and contextual covariates. The cohort commenced with 1927 parent-child dyads comprised of Australian Grade 7 school students, and a parent/guardian. Baseline, one- and two-year follow-up data have been collected, and a three-year follow-up is underway. The data collected include child, familial, parental, and peer factors addressing demographics, alcohol use and supply, parenting practices, other substance use, adolescent behaviours, and peer influences. Baseline data show that only 5.8% of the Grade 7 adolescents had initiated alcohol consumption (of a whole serve of alcohol). Thus, the cohort is ideal for prospectively examining predictors of initiation and progression of alcohol use, which increases markedly through adolescence. Results to date have highlighted the importance of distinguishing between sipping and drinking of full serves of alcohol in the measurement of adolescent alcohol use as these represent distinct behaviours which occur in different environments.

Aims: The aims of this study are to determine if:

1. Parental supply is associated with the progression (acceleration/deceleration) in adolescent drinking over time;
2. The immediate and broader contextual factors mediate or moderate the relationship between parental supply and progression in adolescent drinking over time.

Design: A longitudinal study across three states in Australia (New South Wales, Tasmania, and Western Australia).

Recruitment: Catholic, Independent and Government school in NSW, Tasmania and Western Australia.

Data analysis: Logistic and binomial regression, and multi-level modelling will be used, and latent growth curve modelling (LGCM) within the framework of structural equations modelling (SEM). Moderating and mediating variables, both time variant (e.g., association with alcohol using peers) and time-invariant (e.g. gender) will be modelled. Outcome variables will be modelled using appropriate parametric distributions - Poisson distributions for count data outcomes and binomial distributions for categorical data outcomes. All analyses will be conducted in MPlus v5.2 or Stata. As recommended by Graham imputation of missing data will be done.

Sample size calculations: Due to the flexibility of the modelling approach taken (i.e., the number of parameters allowed to vary), there are a number of different scenarios that can be tested to determine an adequate sample size. The primary interest is in differences in drinking over time between groups who were supplied or not supplied alcohol. Thus, regression analysis will address drinking on a dummy-coded "parental supply" variable. It is hypothesised that parental supply of alcohol would alter the trajectory of harmful drinking by a regression coefficient of ±0.2. This regression coefficient is equivalent to a medium effect size difference between groups, a result which is not unexpected given past research. It was assumed that attrition would result in around 20% missing data on each subsequent measurement occasion. Based on simulation studies, and factoring in potential mediators and moderators, 600 children are required at a minimum. However, as small cell sizes for some associations may affect power, a final sample of ~1800 children and parents has been recruited.

ELIGIBILITY:
Inclusion Criteria:

* Grade 7 High School enrolment
* Parental signed informed consent provided

Exclusion Criteria:

* none

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The cohort includes 1927 Australian adolescents born from 1996-1999 (mean age at baseline: 12.9 years), and a parent or guardian (typically the mother (in 86.3% of dyads; mean age at baseline: 43.9 years)).
Sampling Method: Non-Probability Sample
Enrollment: 1927 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of alcohol consumption | 12 month
  Frequency of alcohol consumption within past 12 months, categorized as: none, 1 day/month, 2-3 days/month, 1 day/week, 2 days/week, 3 days/week, 4 days/week, 5 days/week, 6 days/week, every day.
Typical quantity of alcohol consumption | 12 month
  Quantity of alcohol consumption within past 12 months measured as number of standard drinks (an Australian standard drink contains 10g alcohol).
Frequency of binge drinking | 12 month
  Frequency of drinking more than 4 standard drinks in the past 12 months
Experience of alcohol related harms | 12 months
  17 item scale of alcohol related harms, adapted from the School Health and Alcohol Harm Reduction Project. Scores range from 0 to 85, with higher scores indicating greater experience of harms.
Symptoms of alcohol abuse, dependence and alcohol use disorder | 12 months
  Symptoms of alcohol abuse, dependence, and alcohol use disorder measured via the Diagnostic Interview Schedule for Children 4th Edition. Items correspond to Diagnostic and Statistical Manual of Mental Disorders 4th Edition symptoms of alcohol abuse (4 symptoms), dependence (7 symptoms), and alcohol use disorder (11 symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: RICHARD P MATTICK, PhD, Principal Investigator — NATIONAL DRUG AND ALCOHOL RESEARCH CENTRE, UNSW AUSTRALIA; AMY PEACOCK, PhD, Principal Investigator — NATIONAL DRUG AND ALCOHOL RESEARCH CENTRE, UNSW AUSTRALIA
Locations (1):
- University of New South Wales, Sydney, New South Wales, Australia

REFERENCES:
- [Result] Wadolowski M, Bruno R, Aiken A, Stone C, Najman J, Kypri K, Slade T, Hutchinson D, McBride N, Mattick RP. Sipping, drinking, and early adolescent alcohol consumption: a cautionary note. Alcohol Clin Exp Res. 2015 Feb;39(2):350-4. doi: 10.1111/acer.12613. PMID 25684054
- [Result] Wadolowski M, Hutchinson D, Bruno R, Aiken A, Clare P, Slade T, Najman J, Kypri K, McBride N, Mattick RP. Early Adolescent Alcohol Use: Are Sipping and Drinking Distinct? Alcohol Clin Exp Res. 2015 Sep;39(9):1805-13. doi: 10.1111/acer.12826. Epub 2015 Aug 6. PMID 26248081
- [Result] Wadolowski M, Hutchinson D, Bruno R, Aiken A, Najman JM, Kypri K, Slade T, McBride N, Mattick RP. Parents Who Supply Sips of Alcohol in Early Adolescence: A Prospective Study of Risk Factors. Pediatrics. 2016 Mar;137(3):e20152611. doi: 10.1542/peds.2015-2611. Epub 2016 Feb 26. PMID 26921283
- [Result] Mattick RP, Wadolowski M, Aiken A, Clare PJ, Hutchinson D, Najman J, Slade T, Bruno R, McBride N, Degenhardt L, Kypri K. Parental supply of alcohol and alcohol consumption in adolescence: prospective cohort study. Psychol Med. 2017 Jan;47(2):267-278. doi: 10.1017/S0033291716002373. Epub 2016 Oct 5. PMID 27702422
- [Result] Aiken A, Wadolowski M, Bruno R, Najman J, Kypri K, Slade T, Hutchinson D, McBride N, Mattick RP. Cohort Profile: The Australian Parental Supply of Alcohol Longitudinal Study (APSALS). Int J Epidemiol. 2017 Apr 1;46(2):e6. doi: 10.1093/ije/dyv051. PMID 25953785
- [Result] Aiken A, Clare PJ, Wadolowski M, Hutchinson D, Najman JM, Slade T, Bruno R, McBride N, Kypri K, Mattick RP. Age of Alcohol Initiation and Progression to Binge Drinking in Adolescence: A Prospective Cohort Study. Alcohol Clin Exp Res. 2018 Jan;42(1):100-110. doi: 10.1111/acer.13525. Epub 2017 Nov 21. PMID 29160941
- [Result] Mattick RP, Clare PJ, Aiken A, Wadolowski M, Hutchinson D, Najman J, Slade T, Bruno R, McBride N, Kypri K, Vogl L, Degenhardt L. Association of parental supply of alcohol with adolescent drinking, alcohol-related harms, and alcohol use disorder symptoms: a prospective cohort study. Lancet Public Health. 2018 Feb;3(2):e64-e71. doi: 10.1016/S2468-2667(17)30240-2. Epub 2018 Feb 1. PMID 29396259
- [Result] Sharmin S, Kypri K, Wadolowski M, Bruno R, Khanam M, Aiken A, Hutchinson D, M Najman J, Slade T, McBride N, Attia J, P Mattick R. Parent characteristics associated with approval of their children drinking alcohol from ages 13 to 16 years: prospective cohort study. Aust N Z J Public Health. 2018 Aug;42(4):347-353. doi: 10.1111/1753-6405.12811. Epub 2018 Jul 23. PMID 30035831
- [Result] Sharmin S, Kypri K, Wadolowski M, Bruno R, Khanam M, Aiken A, Hutchinson D, Najman JM, Slade T, McBride N, Attia J, Palazzi K, Oldmeadow C, Mattick RP. Parent hazardous drinking and their children's alcohol use in early and mid-adolescence: prospective cohort study. Eur J Public Health. 2019 Aug 1;29(4):736-740. doi: 10.1093/eurpub/ckz029. PMID 30851106
- [Result] Clare PJ, Aiken A, Yuen WS, Peacock A, Boland V, Wadolowski M, Hutchinson D, Najman J, Slade T, Bruno R, McBride N, Degenhardt L, Kypri K, Mattick RP. Parental supply of alcohol as a predictor of adolescent alcohol consumption patterns: A prospective cohort. Drug Alcohol Depend. 2019 Nov 1;204:107529. doi: 10.1016/j.drugalcdep.2019.06.031. Epub 2019 Aug 29. PMID 31494442
- [Result] Clare PJ, Dobbins T, Bruno R, Peacock A, Boland V, Yuen WS, Aiken A, Degenhardt L, Kypri K, Slade T, Hutchinson D, Najman JM, McBride N, Horwood J, McCambridge J, Mattick RP. The overall effect of parental supply of alcohol across adolescence on alcohol-related harms in early adulthood-a prospective cohort study. Addiction. 2020 Oct;115(10):1833-1843. doi: 10.1111/add.15005. Epub 2020 Mar 6. PMID 32034841
- [Result] Boland VC, Clare PJ, Yuen WS, Peacock A, Aiken A, Wadolowski M, Hutchinson D, Najman J, Slade T, Bruno R, McBride N, Degenhardt L, Kypri K, Mattick RP. The association between parental supply of alcohol and supply from other sources to young people: a prospective cohort. Addiction. 2020 Nov;115(11):2140-2147. doi: 10.1111/add.15033. Epub 2020 Mar 24. PMID 32141130
- [Result] Yuen WS, Chan G, Bruno R, Clare P, Mattick R, Aiken A, Boland V, McBride N, McCambridge J, Slade T, Kypri K, Horwood J, Hutchinson D, Najman J, De Torres C, Peacock A. Adolescent Alcohol Use Trajectories: Risk Factors and Adult Outcomes. Pediatrics. 2020 Oct;146(4):e20200440. doi: 10.1542/peds.2020-0440. Epub 2020 Sep 23. PMID 32968030
- [Result] Aiken A, Clare PJ, Boland VC, Degenhardt L, Yuen WS, Hutchinson D, Najman J, McCambridge J, Slade T, McBride N, De Torres C, Wadolowski M, Bruno R, Kypri K, Mattick RP, Peacock A. Parental supply of sips and whole drinks of alcohol to adolescents and associations with binge drinking and alcohol-related harms: A prospective cohort study. Drug Alcohol Depend. 2020 Oct 1;215:108204. doi: 10.1016/j.drugalcdep.2020.108204. Epub 2020 Aug 5. PMID 32871506
- [Result] Yuen WS, Chan G, Bruno R, Clare PJ, Aiken A, Mattick R, Farrell M, Kypri K, Slade T, Hutchinson D, McBride N, McCambridge J, Boland V, Peacock A. Trajectories of alcohol-induced blackouts in adolescence: early risk factors and alcohol use disorder outcomes in early adulthood. Addiction. 2021 Aug;116(8):2039-2048. doi: 10.1111/add.15415. Epub 2021 Feb 1. PMID 33464664
- [Derived] Aiken A, Chan G, Yuen WS, Clare PJ, Hutchinson D, McBride N, Najman JM, McCambridge J, Upton E, Slade T, Boland VC, De Torres C, Bruno R, Kypri K, Wadolowski M, Mattick RP, Peacock A. Trajectories of parental and peer supply of alcohol in adolescence and associations with later alcohol consumption and harms: A prospective cohort study. Drug Alcohol Depend. 2022 Aug 1;237:109533. doi: 10.1016/j.drugalcdep.2022.109533. Epub 2022 Jun 11. PMID 35752023
- [Derived] Najman JM, Clare PJ, Kypri K, Aiken A, Wadolowski M, Hutchinson D, Slade T, Bruno R, Vogl L, Degenhardt L, Mattick RP. Gender differences in the supply of alcohol to adolescent daughters and sons. Am J Drug Alcohol Abuse. 2021 Jul 4;47(4):508-520. doi: 10.1080/00952990.2021.1927066. Epub 2021 Aug 12. PMID 34383569
- See also: NATIONAL DRUG AND ALCOHOL RESEARCH CENTRE, UNSW, WEBSITE — http://ndarc.med.unsw.edu.au/project/can-parents-teach-their-children-drink-alcohol-responsibly-or-one-drop-drop-too-many